CLINICAL TRIAL: NCT05308641
Title: Effectiveness of Radial Extracorporeal Shockwave Therapy in Patients With Chronic Low Back Pain - Randomized Controlled Trial
Brief Title: Effectiveness of Radial Extracorporeal Shockwave Therapy in Patients With Chronic Low Back Pain
Acronym: ShockEffect
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Dr. med. Tobias Lange, MBA, Principal Investigator, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1_1
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: radial shockwave therapy; chronic low back pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- PreviousSurgery(PrevSurg)_YES/rESWT_4000 (Active Comparator): Previous Surgery on degenerative pathology in lumbar spine: YES rESWT: 4000 pulse, 20 Hz
  Interventions: Procedure: radial extracorporeal shockwave therapy_4000_20; Procedure: standard multimodal pain therapy
- PrevSurg_YES/rESWT_500 (Active Comparator): Previous Surgery on degenerative pathology in lumbar spine: YES rESWT: 500 pulse, 2 Hz
  Interventions: Procedure: radial extracorporeal shockwave therapy_500_2; Procedure: standard multimodal pain therapy
- PrevSurg_YES/rESWT_no (Active Comparator): Previous Surgery on degenerative pathology in lumbar spine: YES rESWT: no
  Interventions: Procedure: standard multimodal pain therapy
- PrevSurg_YES/rESWT_deny (Active Comparator): Previous Surgery on degenerative pathology in lumbar spine: YES rESWT: denied
  Interventions: Procedure: standard multimodal pain therapy
- PrevSurg_NO/rESWT_4000 (Active Comparator): Previous Surgery on degenerative pathology in lumbar spine: NO rESWT: 4000 pulse, 20 Hz
  Interventions: Procedure: radial extracorporeal shockwave therapy_4000_20; Procedure: standard multimodal pain therapy
- PrevSurg_NO/rESWT_500 (Active Comparator): Previous Surgery on degenerative pathology in lumbar spine: NO rESWT: 500 pulse, 2 Hz
  Interventions: Procedure: radial extracorporeal shockwave therapy_500_2; Procedure: standard multimodal pain therapy
- PrevSurg_NO/rESWT_no (Active Comparator): Previous Surgery on degenerative pathology in lumbar spine: NO rESWT: no
  Interventions: Procedure: standard multimodal pain therapy
- PrevSurg_NO/rESWT_deny (Active Comparator): Previous Surgery on degenerative pathology in lumbar spine: NO rESWT: denied
  Interventions: Procedure: standard multimodal pain therapy

INTERVENTIONS:
Procedure: radial extracorporeal shockwave therapy_4000_20 — application of radial extracorporeal shockwave therapy (rESWT) with 4000 pulses and 20 Hz
  Arms: PrevSurg_NO/rESWT_4000; PreviousSurgery(PrevSurg)_YES/rESWT_4000
Procedure: radial extracorporeal shockwave therapy_500_2 — application of radial extracorporeal shockwave therapy (rESWT) with 500 pulses and 2 Hz
  Arms: PrevSurg_NO/rESWT_500; PrevSurg_YES/rESWT_500
Procedure: standard multimodal pain therapy — standard multimodal pain therapy

SUMMARY:
Analysis of the effectiveness of radial shock wave therapy as part of a multimodal pain therapy in the inpatient setting. Different therapy protocols are compared in previously non-operated and in previously operated patients.

DETAILED DESCRIPTION:
Radial shock wave therapy is an approved pain therapy procedure that has been used in various degenerative orthopedic diseases for years. There are a few studies on the subject of chronic back pain. Some studies suggest that this method can be used sensibly. A direct comparison of different therapy protocols has not been carried out so far.

As part of inpatient multimodal pain therapy (including infiltration and physiotherapy) in patients with chronic lumbar back pain with or without degenerative surgery in the area of the lumbar spine radial shock wave therapy after a specific protocol is used. Only inpatients will be admitted to the study. All patients are informed verbally and give their written consent. Comprehensive patient information will be provided before the start of the study, handed out and explained as part of the information discussion. There will be 2 groups ((a) patients with previous degenerative surgery in the area of the lumbar spine, (b) patients without such a pre-operation) examined each with 4 sub-groups depending of the different therapy protocols.

ELIGIBILITY:
Inclusion Criteria:

* chronic lumbar back pain of min 3 months duration

Exclusion Criteria:

* radicular pain of higher intensity than chronic low back pain (cLBP)
* new neurologic deficits
* anticoagulant therapy
* new trauma to the lumbar spine
* spine bacterial infection
* spine tumor
* pregnancy
* coagulation disorder
* previous infiltration to the lumbar spine within 6 weeks prior to study inclusion
* fibromyalgia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-09-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-07 (Estimated)

PRIMARY OUTCOMES:
change in Numeric Rating Scale (NRS) | pre-intervention, 2 weeks, 1 month, 3 months, 6 months
  Pain intensity measured by Numeric Rating Scale (NRS)
  - 11-point scale / min. 0 (better outcome) / max. 10 (worse outcome)

SECONDARY OUTCOMES:
change in Oswestry Disability Index (ODI) | pre-intervention, 2 weeks, 1 month, 3 months, 6 months
  Oswestry Disability Index (ODI)
change in European Quality of Life 5 Dimensions (EQ5D) | pre-intervention, 2 weeks, 1 month, 3 months, 6 months
  European Quality of Life 5 Dimensions (EQ5D)
change in Pain Self-Efficacy Questionnaire (PSEQ) | pre-intervention, 2 weeks, 1 month, 3 months, 6 months
  Pain Self-Efficacy Questionnaire (PSEQ)
change in Patient Health Questionnaire-9 (PHQ-9) | pre-intervention, 2 weeks, 1 month, 3 months, 6 months
  Patient Health Questionnaire-9 (PHQ-9)
change in Perseverative Thinking Questionnaire (PTQ) | pre-intervention, 2 weeks, 1 month, 3 months, 6 months
  Perseverative Thinking Questionnaire (PTQ)
change in Patient Specific Functional Scale (PSFS) | pre-intervention, 2 weeks, 1 month, 3 months, 6 months
  Patient Specific Functional Scale (PSFS)
  * five daily important activities are rated on a 11-point scale
  * min. 0 (worse outcome) / max. 10 (better outcome)
change in The World Health Organisation- Five Well-Being Index (WHO-5) | pre-intervention, 2 weeks, 1 month, 3 months, 6 months
  The World Health Organisation- Five Well-Being Index (WHO-5)
change in Big Five Inventory-SocioOeconomicPanel (BFI-S) | pre-intervention, 2 weeks, 1 month, 3 months, 6 months
  Big Five Inventory-SocioOeconomicPanel (BFI-S)
change in Questionnaire Subgroups for Targeted Treatment (STarT-G) | pre-intervention, 2 weeks, 1 month, 3 months, 6 months
  Subgroups for Targeted Treatment (STarT-G)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias L Schulte, Prof, Study Director — Department of Orthopaedics and Trauma Surgery, St. Josef-Hospital, Ruhr-University Bochum
Locations (1):
- Klinik Blankenstein, Hattingen, Germany

REFERENCES:
- [Result] Lange T, Deventer N, Gosheger G, Lampe LP, Bockholt S, Schulze Boevingloh A, Schulte TL. Effectiveness of Radial Extracorporeal Shockwave Therapy in Patients with Acute Low Back Pain-Randomized Controlled Trial. J Clin Med. 2021 Nov 26;10(23):5569. doi: 10.3390/jcm10235569. PMID 34884271
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8658438/pdf/jcm-10-05569.pdf